CLINICAL TRIAL: NCT05145920
Title: Encouraging Positive Parenting Habits Through Digital Media
Acronym: Habite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: D'Or Institute for Research and Education (Other)
Collaborators: Okinawa Institute of Science and Technology Graduate University (Other); Federal University of Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 50214221.6.0000.5249
Record Dates: First submitted 2021-09-27; First posted 2021-12-06 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: ADHD
Keywords: ADHD; Parent Training; Treatment Access
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Open, single-group trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot testing of an education program promoting effective parenting habit (Experimental): Parents will receive a series of 5 short videos via Whatsapp
  Interventions: Behavioral: HabitE (effective parenting habit) program (in Brazilian Portuguese)

INTERVENTIONS:
Behavioral: HabitE (effective parenting habit) program (in Brazilian Portuguese) — Parents who enroll in the program will receive a series of 5 videos (~ 7 minutes each), 1 video at a time, generally every 3 days. Parents will also receive daily written texts, which include implementation tips and an assessment of a target (transition) behavior.

SUMMARY:
This study evaluates the feasibility and preliminary impacts of a new parenting program consisting of a series of educational videos, delivered via a popular texting platform. For this pilot project, the program content is focused on teaching parents strategies to better manage one of the commonly reported challenges that children face, a transition to a non-preferred activity. Parents with young children demonstrating behavior consistent with ADHD and experiencing difficulties with daily transition routines are invited to participate in the study.

DETAILED DESCRIPTION:
This pilot study employs a pre-post, open trial design with the primary aim to investigate the feasibility of delivering parenting educational materials in a highly accessible format, i.e., a widely used texting platform. The training videos demonstrate the applications of antecedent- and reinforcement-based behavior management techniques in a specific situation and encourage parents to build positive parenting habits. The program usability and satisfaction will be assessed through ratings and answers to open-ended questions by participating parents. The study targets parents of children demonstrating symptoms of ADHD. These families frequently experience difficulties managing everyday routines at home, yet the access to psychosocial treatment is limited. The investigators expect parents to engage well in the program delivered via digital media. Based on the existing literature on the effectiveness of behavior parent training delivered in traditional in-person format, a moderate effect size is expected in the pre-post measures of parenting practices and the child target behavior for this study.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children, aged 4-8, who demonstrate behavior symptoms consistent with ADHD symptoms, i.e., at least 4 inattention and/or 4 hyperactivity/impulsivity symptoms (parent-report). The number of symptoms is lower than the diagnostic threshold to include those with emerging problems. No diagnosis will be made or confirmed in the study. Children need to live with the participating parents at least 5 days per week every week.

Exclusion Criteria:

* Parents of children who have received other forms of pharmacological and/or non-pharmacological treatment in the past 3 months. These parents will be asked to wait to receive other forms of treatment until they complete the study participation.

Parents of children demonstrating symptoms consistent with Autism Spectrum Disorder, and those other difficulties (severe learning, mood and anxiety problems and environmental issues [e.g., recent divorce]) that would better explain the child's challenges transition routines.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — 4 years to 8 years (Child)
Enrollment: 27 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Number of videos viewed | 1 month
  The number of videos viewed (minimum 0, maximum 5) to evaluate participant engagement.
Percentage of completed daily ratings | 1 month
  The percentage of completed daily ratings (minimum 0, maximum 17). Parents are asked to provide daily ratings on the degree of success in implementing parenting strategies taught.
Participant satisfaction | 1 month
  The parent-rated satisfaction regarding information presented in the videos. A rating completed after each video viewing using a 4-point scale. Averaged across the ratings completed for the videos viewed. (Minimum 0, maximum 4). Higher scores indicate greater satisfaction.

SECONDARY OUTCOMES:
Parent-rated child's difficulties with daily transitions | 1 month
  The parent-rated child's difficulties with 9 common daily transitions. Ratings completed before and after the intervention using a 3-point scale. Averaged across the ratings completed for the 9 transitions. Higher scores indicate greater difficulties.
Parent-rated child's impairment related to transition difficulties | 1 month
  The parent-rated level of impairment caused by transition difficulties (1 item). Ratings completed before and after the intervention using a 7 point scale. Higher scores indicate greater impairment.
Proactive parenting | 1 month
  Multidimensional Assessment of Parenting Scale (MAPS) Proactive Parenting sub-scale. Parent ratings completed before and after the intervention using a 5-point scale. Average across 6 items. Higher scores indicate more frequent use of proactive parenting strategies.
Use of positive reinforcement | 1 month
  MAPS Positive Reinforcement sub-scale. Parent ratings completed before and after the intervention using a 5-point scale. Average across 4 items. Higher scores indicate more frequent use of positive reinforcement strategies.
Hostility toward child | 1 month
  MAPS Hostility sub-scale. Parent ratings completed before and after the intervention using a 5-point scale. Average across 7 items. Lower scores indicate less frequent use of hostile reactions during parent-child interactions.

OTHER OUTCOMES:
ADHD symptoms | 1 month
  Strengths and Weakness of Attention-Deficit/Hyperactivity Disorder Symptoms and Normal Behavior Scale (SWAN) inattention and hyperactivity/impulsivity symptoms total. Parent ratings completed before and after the intervention using a 7-point scale. Averaged across 18 items. Higher scores indicate ADHD symptoms more frequently observed.
ODD symptoms | 1 month
  SWAN oppositional/defiant symptoms total. Parent ratings completed before and after the intervention using a 7-point scale. Averaged across 8 items. Higher scores indicate ODD symptoms more frequently observed.
Irritability | 1 month
  Affective Reactivity Index (ARI). Parent ratings completed before and after the intervention using a 3-point scale. Averaged across 6 items. Higher scores indicate irritability more frequently observed.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo E Mattos, MD, PhD, Principal Investigator — D'Or Institute for Research and Eduaction
Locations (1):
- D'Or Institute for Research, Rio de Janeiro, Brazil